CLINICAL TRIAL: NCT02005666
Title: A Randomized, Double-blind, Multicentric, Parallel-group, Active and Placebo Controlled, Three Arm Clinical Study to Compare the Efficacy and Safety of Clindamycin Phosphate 1.2% / Benzoyl Peroxide 5% Gel (of Cadila Healthcare Limited, India) Versus DUAC® Gel (of Stiefel Laboratories, USA) Versus Placebo (Vehicle Gel) in the Ratio of 2:2:1 Respectively, in Patients With Acne Vulgaris
Brief Title: To Compare the Efficacy and Safety of Clindamycin Phosphate 1.2% / Benzoyl Peroxide 5% Gel of CHL Versus DUAC® Gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRL/CT/09/11-12
Record Dates: First submitted 2013-11-28; First posted 2013-12-09 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2017-02

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; DUAC; CADILA; CLIANTHA
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate; Benzoyl Peroxide; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Test-Cadila healthcare limited (Experimental): Drug:-Clindamycin Phosphate 1.2% / Benzoyl Peroxide 5% Gel Dosage Form:-Gel Dosage:-Thin Layer/Pea sized Frequency:-Once a day ,every evening Duration:-77 consecutive days
  Interventions: Drug: Clindamycin Phosphate 1.2% / Benzoyl Peroxide 5% Gel
- Reference (Active Comparator): Drug:-DUAC® Gel (of Stiefel Laboratories, USA) Dosage Form:-Gel Dosage:-Thin Layer/Pea sized Frequency:-Once a day ,every evening Duration:-77 consecutive days
  Interventions: Drug: DUAC® Gel
- Placebo (Placebo Comparator): Drug:-Placebo (Vehicle Gel) Dosage Form:-Gel Dosage:-Thin Layer/Pea sized Frequency:-Once a day ,every evening Duration:-77 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clindamycin Phosphate 1.2% / Benzoyl Peroxide 5% Gel — Drug:-1.2% Clindamycin Phosphate/ 5% Benzoyl Peroxide Gel of Cadila healthcare limited Dosage Form:-Gel Dosage:-Thin Layer/Pea sized Frequency:-Once a day ,every evening Duration:-77 consecutive days
  Other Names: 1.2% Clindamycin Phosphate/ 5% Benzoyl Peroxide Gel of CHL
  Arms: Test-Cadila healthcare limited
Drug: DUAC® Gel — Drug:-DUAC® Gel Dosage Form:-Gel Dosage:-Thin Layer/Pea sized Frequency:-Once a day ,every evening Duration:-77 consecutive days
  Other Names: DUAC® Gel (of Stiefel Laboratories
  Arms: Reference
Drug: Placebo — Drug:-Placebo, Dosage Form:-Gel Dosage:-Thin Layer/Pea sized Frequency:-Once a day ,every evening Duration:-77 consecutive days
  Other Names: Placebo (Vehicle Gel)
  Arms: Placebo

SUMMARY:
This is an Randomized, Double-blind, Multicentric, Parallel-group, Active and Placebo Controlled, Three Arm Clinical Study.

The main objective is to evaluate bioequivalence of Test formulation (Clindamycin Phosphate 1.2%/Benzoyl peroxide 5% gel) of Cadila Healthcare with Reference formulation (DUAC® Gel of Stiefel Laboratories)in the ratio of 2:2:1 of Test drug, Reference drug and Placebo respectively.

Total study duration will be for a period of 78 days which includes treatment duration of 77 days.

850 subjects will be enrolled (randomized)as per the inclusion and exclusion criteria mentioned in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of Acne vulgaris
2. On the face, ≥ 25 non-inflammatory lesions (i.e., open and closed comedones) AND ≥ 20 inflammatory lesions (i.e., papules and pustules) AND ≤ 2 nodulocystic lesions (i.e., nodules and cysts).
3. Investigator's Global Assessment (IGA) of acne severity grade 2, 3 OR 4
4. Willing to refrain from use of all other topical acne medications or antibiotics during the 11 week treatment period.
5. If female of childbearing potential, willing to use an acceptable form of birth control during the study.
6. Have used the same brand of make-up for a minimum period of 2 weeks prior to randomization, for subjects who use make-up, and agree to not change make-up brands or types during the study.
7. Willing to provide written informed consent or assent (HIPAA consent/authorization, as applicable)

Exclusion Criteria:

1. Presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis).
2. Patients who have acne conglobata, acne fulminans and secondary acne (e.g.: chloracne and drug induced acne).
3. Excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris. Well trimmed moustaches are allowed.
4. History of hypersensitivity or allergy to benzoyl peroxide or clindamycin and/or any of the study medication ingredients.
5. Patients who have a severe or intense irritation on the Face.
6. Use within 6 months prior to baseline (Randomization) of oral retinoids (e.g. Accutane®) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
7. Use for less than 3 months prior to baseline (Randomization) of estrogens or oral contraceptives; use of such therapy is allowed if it will remain constant throughout the study.
8. Use on the face within 1 month prior to baseline (Randomization) or during the study of: 1) cryodestruction or chemodestruction, 2) dermabrasion, 3) photodynamic therapy, 4) acne surgery, 5) intralesional steroids, or 6) x-ray therapy.
9. Use within 1 month prior to baseline (Randomization) of: 1) spironolactone, 2) systemic steroids, 3) systemic antibiotics, 4) systemic treatment for acne vulgaris (other than oral retinoids, which require a 6-month washout), or 5) systemic anti-inflammatory agents.
10. Use within 2 weeks prior to baseline (Randomization) of: 1) topical steroids, 2) topical retinoids, 3) topical acne treatments including over-the-counter preparations, 4) topical anti-inflammatory agents, 5) medicated cleansers or 6) topical antibiotics.
11. Patients who have had general anesthesia for any reason and patients who have received neuromuscular blocking agents within 14 days prior to study entry (Randomization).
12. Concomitant use of facial product containing glycolic or other acids, masks, washes or soaps containing benzoyl peroxide or salicylic acid, non mild cleansers or moisturizers containing retinol, salicylic or α- or β-hydroxy acids.
13. Concomitant use of mega-doses of certain vitamins (such as vitamin D and vitamin B12), haloperidol, halogens such as iodide and bromide, lithium, hydantoin and phenobarbital.
14. Facial procedures (chemical or laser peel, microdermabrasion, etc.) within the past 2 weeks or during the study.
15. Concomitant use of tanning booths or sunbathing.
16. A significant medical history of or are currently immunocompromised
17. Have any systemic or dermatologic disease that may affect the evaluation of study results.
18. Have a history of regional enteritis, ulcerative colitis, pseudomembranous colitis or antibiotic-associated colitis.
19. Subjects with clinically significant unstable medical disorders, life-threatening disease, or current malignancies.
20. Subjects who engage in activities that involve excessive or prolonged exposure to sunlight.
21. Subjects with History of Alcohol abuse or other drugs of abuse within 2 years prior to Randomization.
22. Female subjects who are breast-feeding or planning to become pregnant.
23. Subjects who have been treated with an investigational drug or investigational device within a period of 30 days prior to study enrollment.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 850 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Dharmesh Domadia, M.D, Study Director — Cliantha Research Limited
Locations (36):
- United States (12):
  - Universal BioPharma Research, Dinuba, California
  - Research Across America, Santa Ana, California
  - Visions Clinical Research, Boynton Beach, Florida
  - Dermatology Research Instititue, Coral Gables, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Dermatology Specialists, Louisville, Kentucky
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - Discover Research, Bryan, Texas
- India (24):
  - Osmania General Hospital, Hyderabad, Andhra Pradesh
  - Gandhi Hospital,, Hyderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andrapradesh
  - NHL Medical College and VS Hospital, Ahmedabad, Gujarat
  - AMC-MET Medical College, Sheth LG General Hospital,, Ahmedabad, Gujarat
  - Sanjeevani Hospital,, Ahmedabad, Gujarat
  - Dept of Dermatology, Leprosy and STI, Civil Hospital and BJ Medical College,, Ahmedabad, Gujarat
  - Dept of Dermatology, BYL Nair Hospital and TN medical college, Dr ALNair Road, Mumbai Central,, Mumbai, Gujarat
  - Department of Dermatology, New Civil Hospital and Government Medical College, Surat, Gujarat
  - Baroda Medical College, Vadodara, Gujarat
  - Dept of Dermatology, Bhagawan Mahaveer Jain Hospital Millers Road,Vasanthnagar -, Bangalore, Karnataka
  - Dept of Dermatology, Kempegowda Institute of Medical Sciences, Bangalore, Karnataka
  - Sapthagiri Hospital,, Bangalore, Karnataka
  - Dept of Skin & STD, JSS Hospital Ramanuja Road, -, Mysore, Karnataka
  - Government Medical Collge, Nagpur, Maharashtra
  - NKP Salve Institute of Medical Siences and Lata Mangeshkar Hospital,, Nagpur, Maharashtra
  - Dr. D Y Patil Hospital and Research Center, Navi Mumbai, Maharashtra
  - Jehangir Clinical Development Center, Pune, Maharashtra
  - Medipoint Hosp, Pune, Maharashtra
  - Maulana Azad Medical College, New Delhi, National Capital Territory of Delhi
  - Postgraduate Institute of Medical Education & Research (PGIMER), Chandigarh, Punjab
  - M.V. Hospital and research Center, Lucknow, Uttar Pradesh
  - Institute of Post graduate medical and Research, Kolkata, West Bengal
  - Ganga Ram Hospital,, Delhi

REFERENCES:
- [Background] Eller MG, Smith RB, Phillips JP. Absorption kinetics of topical clindamycin preparations. Biopharm Drug Dispos. 1989 Sep-Oct;10(5):505-12. doi: 10.1002/bdd.2510100508. PMID 2804254
- [Background] Zouboulis CC, Fischer TC, Wohlrab J, Barnard J, Alio AB. Study of the efficacy, tolerability, and safety of 2 fixed-dose combination gels in the management of acne vulgaris. Cutis. 2009 Oct;84(4):223-9. PMID 19911678
- See also: 1. Feldman S, Careccia RE, Barham KL, et al. Diagnosis and treatment of acne. Am Fam Physician — http://www.aafp.org/afp/2004/0501/p2123.html
- See also: 2. NilFroushzadeh MA, Siadat AH, Baradaran EH, Moradi S. Clindamycin lotion alone versus combination lotion of clindamycin phosphate plus Tretinoin versus combination lotion of clindamycin phosphate plus salicylic acid in the topical treatment of mild to — http://www.bioline.org.br/pdf?dv09082
- See also: Cleocin T® Prescribing Information — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=16509
- See also: Plaisnce KI, Drusano GL, Forrest A, Townsend RJ, Standiford HC. Pharmacokinetic evaluation of two dosage regimens of clindamycin phosphate. Antimicrob Agents Chemother — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC172501
- See also: DUAC® Gel Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2011/050741s019lbl.pdf
- See also: U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research. Draft Guidance for Industry: Acne Vulgaris: Developing Drugs for Treatment. — http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM071292.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Test-Cadila Healthcare Limited: 1.2% Clindamycin Phosphate/ 5% Benzoyl Peroxide Gel of Cadila healthcare limited Dosage Form:-Gel Dosage:-Thin Layer/Pea sized Frequency:-Once a day ,every evening Duration:-77 consecutive days
- Reference-DUAC® Gel: DUAC® Gel Dosage Form:-Gel Dosage:-Thin Layer/Pea sized Frequency:-Once a day ,every evening Duration:-77 consecutive days
- Placebo: Placebo, Dosage Form:-Gel Dosage:-Thin Layer/Pea sized Frequency:-Once a day ,every evening Duration:-77 consecutive days
Period: Overall Study
Arm/Group | Test-Cadila Healthcare Limited | Reference-DUAC® Gel | Placebo
Started | 338 | 343 | 169
Completed | 311 | 299 | 160
Not Completed | 27 | 44 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test-Cadila Healthcare Limited | Reference-DUAC® Gel | Placebo | Total
Number analyzed (Participants) | 338 | 343 | 169 | 850
Age, Customized [Count of Participants; unit: Participants]
  <18 | 86 | 87 | 47 | 220
  18 - 40 | 252 | 256 | 122 | 630
  41 - 65 | 0 | 0 | 0 | 0
  >65 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 186 | 192 | 103 | 481
  Female | 152 | 151 | 66 | 369
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska | 1 | 1 | 1 | 3
  Asian | 240 | 245 | 121 | 606
  Black | 9 | 8 | 1 | 18
  Native Hawaiian or other pacific Islander | 1 | 0 | 1 | 2
  White | 83 | 88 | 45 | 216
  Other | 4 | 1 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 44 | 50 | 23 | 117
  Non Hispanic/Latino | 294 | 293 | 146 | 733

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline to Week 11 (Study Day 77) for Inflammatory (Papules and Pustules) Lesions.
Description: Mean percent change from baseline to week 11 (study Day 77) for inflammatory (papules and pustules) lesions in PP populations. The primary endpoint of the study is mean percent change from baseline to week 11 (study Day 77) in the inflammatory (papules and pustules) lesion count.
  Papule was Inflammatory lesion; small (< 5mm in diameter), solid palpable lesion, usually with inflamed elevation of the skin that does not contain pus. Pustule was Inflammatory lesion; small (< 5mm in diameter), inflamed skin swelling that is filled with pus. The test product was judged therapeutically equivalent to the reference product in the reduction of inflammatory lesions if the 90% confidence interval was contained within the interval (0.80, 1.25)
Time Frame: week 11
Measure: Mean (Standard Deviation); unit: percentage of mean change from baseline
Arm/Group | Test-Cadila Healthcare Limited | Reference-DUAC® Gel | Placebo
Number analyzed (Participants) | 236 | 233 | 128
percentage of mean change from baseline | -67.6 (28.39) | -71.3 (25.98) | -51.9 (33.99)

2. Secondary Outcome: Mean Percent Change From Baseline to Week 11 in the Non-inflammatory Lesion Count
Description: Mean percent change from baseline to week 11 in the non-inflammatory lesion count. The mean percent change from baseline to week 11 in the non-inflammatory (open and closed comedones) lesion count in per protocol population . The analysis was same as the analysis performed for the mean percent reduction from baseline to Day 77 in the number of inflammatory lesion count.
  Closed Comedone was Non-inflammatory lesion; whitehead, skin-colored or slightly inflamed "bump" in the skin. Open Comedone was Non-inflammatory lesion; blackhead, surface of the plugged sebaceous follicle has a blackish appearance. The test product was judged therapeutically equivalent to the reference product in the reduction of Non inflammatory lesions if the 90% confidence interval was contained within the interval (0.80, 1.25)
Time Frame: week 11
Population: Total randomized subjects 850,in 2:2:1 ratio(Test:338,Reference:343,Placebo:169).80 subjects withdrawn,770 subjects completed study.Efficacy analysis done in Per Protocol (PP)Population, total 253 subjects were excluded from total randomized subjects.For efficacy analysis,597 subjects considered in PP population (Test:236,Reference:233,Placebo:128)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Test-Cadila Healthcare Limited | Reference-DUAC® Gel | Placebo
Number analyzed (Participants) | 236 | 233 | 128
percentage of change | -61.7 (29.50) | -61.3 (28.46) | -42.0 (34.99)

3. Secondary Outcome: Proportion of Subjects With a Clinical Response of "Success" at Week 11
Description: Success was defined as an Investigator Global Assessment (IGA) score that is at least 2 grades less than the baseline assessment.
  Percentage of subjects with at least 2 grades improvement in IGA scoring from baseline to week 11 for test, reference and placebo in Per protocol population.
  IGA is evaluated in the range of 0 to 4. Grade 0=Clear skin with no inflammatory or non-inflammatory lesions;Grade 1=Almost clear;rare non-inflammatory lesions with no more than one small inflammatory lesion; Grade 2 = Mild severity; greater than grade 1;some non-inflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions);Grade 3 = Moderate severity; greater than Grade 2; up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion;Grade 4= Severe; greater than Grade 3;up to many non-inflammatory lesions and may have some inflammatory lesions,but no more than a few nodular lesions
Time Frame: Week 11
Measure: Count of Participants; unit: Participants
Arm/Group | Test-Cadila Healthcare Limited | Reference-DUAC® Gel | Placebo
Number analyzed (Participants) | 236 | 233 | 128
Participants
  Success Rate | 40 | 32 | 10
  Failure Rate | 196 | 201 | 118

ADVERSE EVENTS:
Time Frame: Day 1 to Day 78
Groups:
- Test-Cadila Healthcare Limited: 1.2% Clindamycin Phosphate/ 5% Benzoyl Peroxide Gel of Cadila healthcare limited Dosage Form:-Gel Dosage:-Thin Layer/Pea sized Frequency:-Once a day ,every evening Duration:-77 consecutive days Other Name: 1.2% Clindamycin Phosphate/ 5%
Arm/Group | Test-Cadila Healthcare Limited | Reference-DUAC® Gel | Placebo
All-Cause Mortality (participants affected / at risk) | 0/338 | 0/343 | 0/169
Serious Adverse Events (participants affected / at risk) | 0/338 | 0/343 | 0/169
Other Adverse Events (participants affected / at risk) | 59/338 | 61/343 | 29/169
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test-Cadila Healthcare Limited (N=338) | Reference-DUAC® Gel (N=343) | Placebo (N=169)
Application site dryness (General disorders) | 7 (7) | 7 (7) | 2 (2)
Application site erythema (General disorders) | 2 (2) | 2 (2) | 4 (4)
Application site oedema (General disorders) | 1 (1) | 1 (1) | 1 (1)
Application site pain (General disorders) | 2 (2) | 3 (3) | 2 (2)
Application site pruritus (General disorders) | 2 (2) | 4 (4) | 3 (3)
Facial pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (11) | 10 (10) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 9 (9) | 15 (15) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Scleral cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Ear deformity acquired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes